CLINICAL TRIAL: NCT03677141
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized, Controlled Study Investigating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Mosunetuzumab (BTCT4465A) in Combination With CHOP or CHP-Polatuzumab Vedotin in Patients With B-Cell Non-Hodgkin Lymphoma
Brief Title: A Phase Ib/II Study Investigating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Mosunetuzumab (BTCT4465A) in Combination With CHOP or CHP-Polatuzumab Vedotin in Participants With B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO40515; 2018-001039-29 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — polatuzumab vedotin; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase Ib: Mosunetuzumab (M)-CHOP Dose Finding (Experimental): Participants will receive M-CHOP up to the phase II recommended dose (RP2D).
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Tocilizumab
- Phase Ib: M-CHP-Pola Dose-Finding (Experimental): Participants will receive M-CHP-Pola up to the RP2D.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Tocilizumab
- Phase II: M-CHOP Previously Untreated (1L) DLBCL Safety Cohort (Experimental): Participants with 1L DLBCL will receive mosunetuzumab at the RP2D in combination with CHOP.
  Interventions: Drug: Mosunetuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Tocilizumab
- Phase II: M-CHP-Pola 1L DLBCL (Experimental): Participants with 1L DLBCL will receive M-CHP-Pola at a dose determined in the dose finding stage.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Tocilizumab
- Phase II: Rituxumab (R)-CHP-Pola 1L DLBCL (Active Comparator): Participants with 1L DLBCL will receive R-CHP-Pola at a dose determined in the dose finding stage.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituxumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone
- Phase II: M-CHOP 1L DLBCL (Experimental): Participants with 1L DLBCL will receive M-CHOP at a dose determined in the dose finding stage.
  NOTE: No participants were enrolled to this arm.
  Interventions: Drug: Mosunetuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Tocilizumab

INTERVENTIONS:
Drug: Mosunetuzumab — Participants will receive intravenous (IV) mosunetuzumab.
  Arms: Phase II: M-CHOP 1L DLBCL; Phase II: M-CHOP Previously Untreated (1L) DLBCL Safety Cohort; Phase II: M-CHP-Pola 1L DLBCL; Phase Ib: M-CHP-Pola Dose-Finding; Phase Ib: Mosunetuzumab (M)-CHOP Dose Finding
Drug: Polatuzumab Vedotin — Participants will receive polatuzumab vedotin via IV.
  Arms: Phase II: M-CHP-Pola 1L DLBCL; Phase II: Rituxumab (R)-CHP-Pola 1L DLBCL; Phase Ib: M-CHP-Pola Dose-Finding; Phase Ib: Mosunetuzumab (M)-CHOP Dose Finding
Drug: Rituxumab — Participants will receive rituxumab via IV.
  Arms: Phase II: Rituxumab (R)-CHP-Pola 1L DLBCL
Drug: Cyclophosphamide — Participants will receive cyclophosphamide via IV.
Drug: Doxorubicin — Participants will receive doxorubicin via IV.
Drug: Vincristine — Participants will receive vincristine via IV.
  Arms: Phase II: M-CHOP 1L DLBCL; Phase II: M-CHOP Previously Untreated (1L) DLBCL Safety Cohort; Phase Ib: Mosunetuzumab (M)-CHOP Dose Finding
Drug: Prednisone — Participants will receive oral prednisone.
Drug: Tocilizumab — Participants will receive tocilizumab via IV.
  Arms: Phase II: M-CHOP 1L DLBCL; Phase II: M-CHOP Previously Untreated (1L) DLBCL Safety Cohort; Phase II: M-CHP-Pola 1L DLBCL; Phase Ib: M-CHP-Pola Dose-Finding; Phase Ib: Mosunetuzumab (M)-CHOP Dose Finding

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and preliminary efficacy of mosunetuzumab in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone (M-CHOP) and, subsequently, in combination with cyclophosphamide, doxorubicin, and prednisone (CHP) plus polatuzumab vedotin (CHP-pola) in participants with relapsed or refractory (R/R) B-cell non-Hodgkin lymphoma (NHL), and in previously untreated participants with diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria for Phase Ib and Phase II Portions

* At least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest diameter
* Eastern Cooperative Oncology Group Performance Status of 0, 1, or 2
* Adequate hematologic function

Inclusion Criteria for Phase Ib Portion

Participants must also meet the following criteria for study entry into the Phase Ib portion:

* Histologically confirmed B-cell NHL according to the World Health Organization (WHO) 2016 classification expected to express the cluster of differentiation-20 (CD20) antigen
* Relapsed or refractory (R/R) B-cell NHL after at least one prior systemic lymphoma therapy
* Treatment with at least one prior CD20-directed therapy
* Group B only: no prior treatment with polatuzumab vedotin

Inclusion Criteria for Phase II Portion

Participants must also meet the following criteria for study entry in the Phase II portion:

* Previously untreated, histologically confirmed DLBCL according to WHO 2016 classification
* International Prognostic Index (IPI) score of 2-5

Exclusion Criteria

* Prior treatment with mosunetuzumab
* Prior allogenic stem-cell transplant
* Current Grade >1 peripheral neuropathy
* Participants with history of confirmed progressive multifocal leukoencephalopathy (PML)
* Known or suspected chronic active Epstein Barr virus (CAEBV), hepatitis B, hepatitis C (HCV), or Human Immunodeficiency Virus (HIV)
* Prior solid organ transplantation
* History of autoimmune disease
* Current or past history of central nervous system (CNS) lymphoma
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Significant cardiovascular disease or pulmonary disease
* Clinically significant history of liver disease
* Recent major surgery within 4 weeks before the start of C1D1, other than superficial lymph node biopsies for diagnosis

Exclusion Criteria for Phase Ib Portion

Participants who also meet any of the following criteria will be excluded from study entry in the Phase Ib portion:

* Prior treatment with chemotherapy, immunotherapy, and biologic therapy 4 weeks prior to C1D1
* Prior treatment with radiotherapy within 2 weeks prior to C1D1
* Adverse events from prior anti-cancer therapy resolved to ≤Grade 1 (with the exception of alopecia and anorexia)
* Prior treatment with >250 mg/m^2 doxorubicin (or equivalent anthracycline dose)

Exclusion Criteria for Phase II Portion

Participants who also meet any of the following criteria will be excluded from study entry in the Phase II portion:

* Participants with transformed lymphoma
* Prior therapy for B-cell NHL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (15):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of California; Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles (UCLA) - Hematology/Oncology Santa Monica, Santa Monica, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Scott and White Hospital; Cancer Center, Temple, Texas
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Austria (4):
  - Uniklinikum Salzburg, LKH; Univ.Klinik f. Innere Medizin III der PMU, Salzburg
  - LKH Steyr, Steyr
  - Medizinische Universität Wien, Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Hanusch-Krankenhaus, Vienna
- France (5):
  - CHU Henri Mondor; Service d'Oncologie Medicale, Créteil
  - Centre Leon Berard, Lyon
  - Hôpital Saint-Louis, Paris
  - Centre Henri Becquerel- Centre de Lutte Contre le Cancer, Saint-Herblain
  - Gustave Roussy, Villejuif
- Poland (5):
  - Maria Sklodowska-Curie Memorial Cancer Centre, Gliwice
  - Ma?opolskie Centrum Medyczne, Krakow
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka, Słupsk
  - Instytut Hematologii i Transfuzjologii; Klinika Zaburze? Hemostazy i Chorób Wewn?trznych, Warsaw
  - Katedra i Klinika Hematologii; Nowotworów Krwi i Transplantacji Szpiku, Wroc?aw
- South Korea (4):
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcantara; Servicio de Hematología, Cáceres
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Westin J, Phillips TJ, Mehta A, Hoffmann MS, Gonzalez-Barca E, Thieblemont C, Bastos-Oreiro M, Greil R, Giebel S, Wei MC, Wang J, Bucher R, Sit J, Penuel E, Purev E, Yee DL, Bergua-Burgues JM. Mosunetuzumab plus Pola-CHP compared with Pola-R-CHP in previously untreated DLBCL: final results from a phase 2 study. Blood Adv. 2025 May 27;9(10):2461-2472. doi: 10.1182/bloodadvances.2024014907. PMID 39908481
- [Derived] Olszewski AJ, Phillips TJ, Hoffmann MS, Armand P, Kim TM, Yoon DH, Mehta A, Greil R, Westin J, Lossos IS, Munoz JL, Sit J, Wei MC, Yang A, Chen V, Purev E, Yee DL, Jaeger U. Mosunetuzumab in combination with CHOP in previously untreated DLBCL: safety and efficacy results from a phase 2 study. Blood Adv. 2023 Oct 24;7(20):6055-6065. doi: 10.1182/bloodadvances.2023010840. PMID 37581593

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A1: Phase Ib Mosunetuzumab + CHOP: Participants with relapsed/refractory (R/R) B-cell non-Hodgkin lymphoma (NHL) received mosunetuzumab on Cycle 1 Day 1 (C1D1), C1D8, and C1D15, then on Day 1 of subsequent cycles. In addition, participants received cyclophosphamide, doxorubicin, and vincristine on D1, and prednisone on D1-D5 (CHOP). Treatment was given for 6 cycles (cycle length = 21 days).
- Group A2: Phase Ib Mosunetuzumab + CHOP: Participants with relapsed/refractory (R/R) B-cell NHL received mosunetuzumab on Cycle 1 Day 1 (C1D1), C1D8, and C1D15, then on Day 1 of subsequent cycles. In addition, participants received cyclophosphamide, doxorubicin, and vincristine on D1, and prednisone on D1-D5. Treatment was given for 6 cycles (cycle length = 21 days).
- Group B: Phase Ib Mosunetuzumab + CHP-Pola: Participants with R/R NHL received 6 cycles of mosunetuzumab (M) + cyclophosphamide, doxorubicin, prednisone (CHP), and polatuzumab vedotin (Pola) (cycle length = 21 days). Participants received M on C1D2, C1D8, C1D15, C2D2, and on D1 of subsequent cycles if well tolerated. CHP-pola was given on D1 of each cycle (D1-D5 for prednisone).
- Group C: Phase II Mosunetuzumab + CHOP: Participants with previously untreated diffuse large B-cell lymphoma (DLBCL) received mosunetuzumab on Cycle 1 Day 1 (C1D1), C1D8, and C1D15, then on Day 1 of subsequent cycles. In addition, participants received cyclophosphamide, doxorubicin, and vincristine on D1, and prednisone on D1-D5 (CHOP). Treatment was given for 6 cycles (cycle length = 21 days).
- Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized): Participants received M-CHP-Pola for 6 cycles (cycle length = 21 days). Participants received M on C1D1, C1D8, and C1D15, then on D1 of subsequent cycles. CHP-pola was given on D1 of each cycle (D1-D5 for prednisone).
- Arm 2: Phase II Rituximab + CHP-Pola (Randomized): Participants received R-CHP-Pola for 6 cycles (cycle length = 21 days). R-CHP-pola was given on D1 of each cycle (D1-D5 for prednisone).
Period: Overall Study
Arm/Group | Group A1: Phase Ib Mosunetuzumab + CHOP | Group A2: Phase Ib Mosunetuzumab + CHOP | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Started | 3 | 4 | 8 | 40 | 40 | 22
Completed | 1 | 3 | 1 | 28 | 31 | 19
Not Completed | 2 | 1 | 7 | 12 | 9 | 3
Not completed — Death | 2 | 1 | 6 | 9 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Screen failure or enrolled in error | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A1: Phase Ib Mosunetuzumab + CHOP | Group A2: Phase Ib Mosunetuzumab + CHOP | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized) | Total
Number analyzed (Participants) | 3 | 4 | 8 | 40 | 40 | 22 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.0 (13.0) | 71.3 (3.4) | 60.1 (18.0) | 63.4 (11.0) | 65.0 (10.0) | 57.7 (14.3) | 63.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 18 | 14 | 8 | 44
  Male | 3 | 3 | 5 | 22 | 26 | 14 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 3 | 2 | 3 | 12
  Not Hispanic or Latino | 3 | 3 | 5 | 36 | 35 | 18 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 10 | 5 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 4 | 8 | 28 | 30 | 20 | 93
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 4 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate at the Time of Primary Response Assessment (PRA) Based on Positron Emission Tomography - Computed Tomography (PET-CT) as Determined by Independent Review Committee (IRC)
Description: The CR rate was defined as the percentage of participants with CR. Assessments were made according to the Lugano 2014 Response Criteria.
Time Frame: 6-8 weeks after either C6D1 or last dose of study treatment
Population: The intent-to-treat (ITT) population consisted of all participants. Efficacy analyses for Arms A1, A2, and B were exploratory. The primary efficacy analysis compared Arm 1 vs Arm 2, with participants grouped according to the treatment arm assigned at randomization. Group C was included in secondary efficacy analysis, and efficacy analyses for Arms A1, A2, and B were exploratory.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 22
Percentage of participants | 72.5 [56.11 to 85.40] | 77.3 [54.63 to 92.18]
Statistical Analysis 1: Comparison: Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) vs Arm 2: Phase II Rituximab + CHP-Pola (Randomized); Test type: Superiority; Difference in rates = -4.77, 95% CI 2-sided [-30.61 to 21.07]

2. Secondary Outcome: CR Rate at PRA Based on CT Only as Determined by the Investigator (Phase II)
Time Frame: 6-8 weeks after C6D1 or last dose of study treatment
Population: The intent-to-treat (ITT) population consisted of all participants. Efficacy analyses for Arms A1, A2, and B were exploratory.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 40 | 22
Percentage of participants | 50.0 [33.80 to 66.20] | 47.5 [31.51 to 63.87] | 31.8 [13.86 to 54.87]

3. Secondary Outcome: Overall Response Rate (ORR) at PRA Based on PET-CT as Determined by the Investigator (Phase II)
Description: ORR is defined as a CR or PR at the time of primary assessment based on PET-CT, as determined by the investigator.
Time Frame: 6-8 weeks after C6D1 or last dose of study treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 40 | 22
Percentage of participants | 87.5 [73.20 to 95.81] | 80.0 [64.35 to 90.95] | 77.3 [54.63 to 92.18]

4. Secondary Outcome: ORR at PRA Based on CT Only as Determined by the Investigator (Phase II)
Description: ORR is defined as a CR or PR at the time of primary assessment based on CT only, as determined by the investigator.
Time Frame: 6-8 weeks after C6D1 or last dose of study treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 40 | 22
Percentage of participants | 85.0 [70.16 to 94.29] | 72.5 [56.11 to 85.40] | 81.8 [59.72 to 94.81]

5. Secondary Outcome: Best ORR Based on PET-CT and/or CT Scan as Determined by the Investigator (Phase II)
Description: Best ORR was defined as CR or PR at any time on study and based on PET-CT or CT only as determined by the investigator.
Time Frame: Up to approximately 50 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 36 | 22
Percentage of responders | 95.0 [83.08 to 99.39] | 85.0 [70.16 to 94.29] | 95.5 [77.16 to 99.88]

6. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator (Phase II)
Description: DOR is defined as the time from the first occurrence of a documented objective response to disease progression or relapse as determined by the investigator, or death from any cause, whichever occurs first. The range values (min-max) are based on censored observations (if a participant did not experience disease progression or death prior to the end of the trial DOR was censored on the date of the last tumor assessment).
Time Frame: Up to approximately 50 months
Population: The number of participants analyzed was the number of participants with a PR or CR in each arm. The range values (min-max) are based on censored observations (if a participant did not experience disease progression or death prior to the end of the trial DOR was censored on the date of the last tumor assessment). Efficacy analyses for Arms A1, A2, and B were exploratory.
Measure: Median (Full Range); unit: Months
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 38 | 34 | 21
Months | NA [0 to 28] — This value could not be determined due to an insufficient number of participants with the event. | NA [0 to 28] — This value could not be determined due to an insufficient number of participants with the event. | NA [1 to 27] — This value could not be determined due to an insufficient number of participants with the event.

7. Secondary Outcome: Progression-free Survival (PFS) as Determined by the Investigator (Phase II)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression or relapse as determined by the investigator, or death from any cause, whichever occurs first. The earliest contributing event to PFS is reported. The range (min-max) values are based on censored observations (participants without a baseline-evaluable tumor assessment were censored at the date of randomization or first study treatment, plus 1 day).
Time Frame: Up to approximately 50 months
Population: Efficacy analyses for Arms A1, A2, and B were exploratory. The number of participants analyzed reflects the number of participants with the event. The range (min-max) values are based on censored observations (participants without a baseline-evaluable tumor assessment were censored at the date of randomization or first study treatment, plus 1 day).
Measure: Median (Full Range); unit: Months
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 40 | 22
Months | NA [0 to 31] — This value could not be determined due to an insufficient number of participants with the event. | NA [0 to 30] — This value could not be determined due to an insufficient number of participants with the event. | NA [3 to 30] — This value could not be determined due to an insufficient number of participants with the event.

8. Secondary Outcome: PFS at 1 Year as Determined by the Investigator (Phase II)
Description: PFS at 1 year is defined as the proportion of participants with disease progression or relapse as determined by the investigator, or death from any cause within 1 year of randomization.
Time Frame: 1 year
Population: Efficacy analyses for Arms A1, A2, and B were exploratory.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 40 | 22
Percentage of participants | 77.47 [63.65 to 91.29] | 70.83 [55.59 to 86.07] | 81.82 [65.70 to 97.94]

9. Secondary Outcome: Event-free Survival (EFS) as Determined by the Investigator (Phase II)
Description: EFS is defined as the time from randomization to the first occurrence of disease progression or relapse, as determined by the investigator, initiation of new anti-lymphoma therapy (NALT), or death from any cause, whichever occurs first. The range values (min-max) are based on censored observations (if a participant did not experience disease progression or death prior to the end of the trial DOR was censored on the date of the last tumor assessment).
Time Frame: Up to 50 months
Population: Efficacy analyses for Arms A1, A2, and B were exploratory. The number of participants analyzed reflects the number of participants with the event. The range (min-max) values are based on censored observations (participants without a baseline-evaluable tumor assessment or documentation of NALT were censored at the date of randomization or first study treatment, plus 1 day).
Measure: Median (Full Range); unit: Months
Arm/Group | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 12 | 11 | 5
Months | NA [2 to 31] — This value could not be determined due to an insufficient number of participants with the event. | NA [0 to 30] — This value could not be determined due to an insufficient number of participants with the event. | NA [3 to 30] — This value could not be determined due to an insufficient number of participants with the event.

10. Secondary Outcome: Time to Deterioration in Lymphoma Symptoms as Measured by the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Subscale
Time Frame: C1D1 through follow-up period (to begin 2 years after PRA or at the time of study drug discontinuation)
Population: The intent-to-treat (ITT) population consisted of all participants. Efficacy analyses for Arms A1, A2, and B were exploratory. Patient-reported outcomes (PROs) were evaluated only for Arm 1 and Arm 2 per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 22
Months | NA [2.3 to NA] — Value was not estimable due to an insufficient number of participants with the event. | 6.5 [2.1 to NA] — Value was not estimable due to an insufficient number of participants with the event.

11. Secondary Outcome: Time to Deterioration in Physical Functioning and Fatigue as Measured by the European Organization for Research and Treatment of Cancer Quality of Life - Core 30 Questionnaire (EORTC QLQ-C30)
Time Frame: C1D1 through follow-up period (to begin 2 years after PRA or at the time of study drug discontinuation)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 40 | 22
Months | 2.3 [1.2 to 5.4] | 2.3 [0.8 to NA] — Value was not estimable due to an insufficient number of participants with the event.

12. Secondary Outcome: Polatuzumab Vedotin Serum Concentrations
Time Frame: C2D1, C6D1
Population: Participants with at least one pharmacokinetic (PK) sample were included in analysis. Arms in which participants did not receive polatuzumab vedotin were not included in this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 8 | 40 | 22
ug/mL
  C2D1 pre-dose: number analyzed (Participants) | 6 | 33 | 18
  C2D1 pre-dose | 0.993 (779.4) | 1.99 (80.7) | 1.73 (107.9)
  C6D1 pre-dose: number analyzed (Participants) | 4 | 27 | 20
  C6D1 pre-dose | 2.76 (820.1) | 8.13 (34.5) | 5.8 (42)

13. Secondary Outcome: Polatuzumab Vedotin Antibody-conjugated Monomethyl Auristatin E (acMMAE) Serum Concentrations
Time Frame: C1D1-C6D1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 8 | 40 | 22
ng/mL
  C1D1 post-dose: number analyzed (Participants) | 8 | 22 | 16
  C1D1 post-dose | 620 (54.5) | 668 (21.2) | 584 (23.1)
  C1D2 pre-dose: number analyzed (Participants) | 7 | 0 | 0
  C1D2 pre-dose | 219 (412.2) |  |
  C1D2 24hrs post-dose: number analyzed (Participants) | 8 | 24 | 0
  C1D2 24hrs post-dose | 115 (658.3) | 275 (28.2) |
  C1D8 pre-dose: number analyzed (Participants) | 7 | 29 | 0
  C1D8 pre-dose | 23 (1040.4) | 42 (82) |
  C1D15 pre-dose: number analyzed (Participants) | 7 | 30 | 0
  C1D15 pre-dose | 8.22 (550.4) | 13.2 (87.4) |
  C2D1 pre-dose: number analyzed (Participants) | 6 | 31 | 18
  C2D1 pre-dose | 4.87 (626) | 6.81 (80.1) | 7.09 (95.5)
  C2D1 post-dose: number analyzed (Participants) | 6 | 32 | 13
  C2D1 post-dose | 656 (21.1) | 653 (18) | 654 (21)
  C3D1 pre-dose: number analyzed (Participants) | 5 | 33 | 0
  C3D1 pre-dose | 19.2 (58.7) | 15.8 (39.5) |
  C3D1 post-dose: number analyzed (Participants) | 5 | 30 | 0
  C3D1 post-dose | 144 (112947.3) | 544 (90.7) |
  C4D1 pre-dose: number analyzed (Participants) | 4 | 33 | 21
  C4D1 pre-dose | 16.8 (79.6) | 16.8 (50.3) | 15.6 (41.4)
  C4D1 post-dose: number analyzed (Participants) | 4 | 30 | 18
  C4D1 post-dose | 783 (26.5) | 614 (15.4) | 696 (24.1)
  C5D1 pre-dose: number analyzed (Participants) | 3 | 29 | 0
  C5D1 pre-dose | 7.14 (343.5) | 19 (39.7) |
  C5D1 post-dose: number analyzed (Participants) | 3 | 9 | 0
  C5D1 post-dose | 544 (37.6) | 605 (21.6) |
  C6D1 pre-dose: number analyzed (Participants) | 4 | 25 | 19
  C6D1 pre-dose | 11.8 (476.6) | 21.2 (34.7) | 17.3 (40.8)

14. Secondary Outcome: Polatuzumab Vedotin Unconjugated Mono-methyl Auristatin E (MMAE) Serum Concentrations
Time Frame: C1D1-C6D1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 8 | 40 | 22
ng/mL
  C1D1 post-dose: number analyzed (Participants) | 8 | 29 | 16
  C1D1 post-dose | 0.535 (464.6) | 0.55 (71.1) | 0.432 (78.8)
  C1D2 pre-dose: number analyzed (Participants) | 7 | 0 | 0
  C1D2 pre-dose | 1.94 (114.2) |  |
  C1D2 24hrs post-dose: number analyzed (Participants) | 8 | 30 | 0
  C1D2 24hrs post-dose | 3.3 (97.8) | 2.82 (51.9) |
  C1D8 pre-dose: number analyzed (Participants) | 7 | 30 | 0
  C1D8 pre-dose | 2.95 (80.9) | 1.27 (93.6) |
  C1D15 pre-dose: number analyzed (Participants) | 7 | 30 | 0
  C1D15 pre-dose | 0.604 (113.3) | 0.301 (104.1) |
  C2D1 pre-dose: number analyzed (Participants) | 6 | 33 | 18
  C2D1 pre-dose | 0.187 (47.3) | 0.0773 (110.2) | 0.0697 (87)
  C2D1 post-dose: number analyzed (Participants) | 6 | 35 | 14
  C2D1 post-dose | 0.238 (64) | 0.137 (84) | 0.116 (56.3)
  C3D1 pre-dose: number analyzed (Participants) | 5 | 33 | 0
  C3D1 pre-dose | 0.168 (92) | 0.146 (96.9) |
  C3D1 post-dose: number analyzed (Participants) | 5 | 32 | 0
  C3D1 post-dose | 0.111 (173.9) | 0.203 (92.7) |
  C4D1 pre-dose: number analyzed (Participants) | 4 | 33 | 21
  C4D1 pre-dose | 0.0491 (NA) — If more than one-third of values were lower than reportable, only the median, maximum, and geometric mean are reported. | 0.14 (93.8) | 0.106 (88.9)
  C4D1 post-dose: number analyzed (Participants) | 4 | 30 | 18
  C4D1 post-dose | 0.0825 (188.3) | 0.186 (66.1) | 0.164 (43.6)
  C5D1 pre-dose: number analyzed (Participants) | 3 | 30 | 0
  C5D1 pre-dose | 0.0741 (247) | 0.137 (74.4) |
  C5D1 post-dose: number analyzed (Participants) | 3 | 7 | 0
  C5D1 post-dose | 0.212 (54.2) | 0.17 (38.1) |
  C6D1 pre-dose: number analyzed (Participants) | 4 | 27 | 19
  C6D1 pre-dose | 0.0967 (194.2) | 0.142 (63.8) | 0.0974 (82.4)

15. Secondary Outcome: Mosunetuzumab Serum Concentrations
Time Frame: C1D1-C5D1
Population: Participants with at least one pharmacokinetic (PK) sample were included in analysis. Arms in which participants did not receive mosunetuzumab were not included in this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Group A1: Phase Ib Mosunetuzumab + CHOP | Group A2: Phase Ib Mosunetuzumab + CHOP | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized)
Number analyzed (Participants) | 3 | 4 | 8 | 40 | 40
ug/mL
  C1D1 post-dose: number analyzed (Participants) | 3 | 4 | 0 | 37 | 22
  C1D1 post-dose | 0.157 (22.1) | 0.181 (26.7) |  | 0.155 (34.1) | 0.132 (73.2)
  C1D1 2 hrs post-dose: number analyzed (Participants) | 3 | 4 | 0 | 35 | 0
  C1D1 2 hrs post-dose | 0.152 (27.8) | 0.163 (25.8) |  | 0.151 (28.1) |
  C1D2 2 hrs post-dose: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0
  C1D2 2 hrs post-dose |  |  | 0.145 (80) |  |
  C1D2 24 hrs post-dose: number analyzed (Participants) | 3 | 4 | 8 | 36 | 29
  C1D2 24 hrs post-dose | 0.103 (23.3) | 0.112 (8.1) | 0.0947 (60.2) | 0.096 (35.7) | 0.0825 (46.1)
  C1D8 pre-dose: number analyzed (Participants) | 3 | 3 | 7 | 39 | 35
  C1D8 pre-dose | 0.0331 (49) | 0.0218 (153.2) | 0.0334 (113.6) | 0.0253 (62.2) | 0.0263 (77)
  C1D8 post-dose: number analyzed (Participants) | 3 | 3 | 7 | 39 | 35
  C1D8 post-dose | 0.342 (18.8) | 0.427 (36.2) | 0.354 (36.9) | 0.426 (30.3) | 0.376 (38.8)
  C1D8 2hrs post-dose: number analyzed (Participants) | 3 | 4 | 7 | 38 | 0
  C1D8 2hrs post-dose | 0.32 (28.5) | 0.409 (50.1) | 0.349 (43.1) | 0.388 (27.6) |
  C1D15 pre-dose: number analyzed (Participants) | 3 | 4 | 7 | 39 | 31
  C1D15 pre-dose | 0.0866 (47.9) | 0.0884 (52.8) | 0.0911 (57.7) | 0.0953 (41.8) | 0.102 (47.7)
  C1D15 post-dose: number analyzed (Participants) | 3 | 4 | 7 | 39 | 31
  C1D15 post-dose | 2.83 (22.6) | 5.71 (38.6) | 5.72 (44) | 7.13 (27.7) | 6.31 (34.8)
  C1D15 2 hrs post-dose: number analyzed (Participants) | 2 | 4 | 7 | 38 | 0
  C1D15 2 hrs post-dose | 2.28 (7.5) | 5.66 (38.7) | 5.92 (18.5) | 6.56 (28.4) |
  C2D1 pre-dose: number analyzed (Participants) | 2 | 4 | 0 | 37 | 33
  C2D1 pre-dose | 0.549 (24.3) | 1.52 (49.4) |  | 1.67 (32.1) | 1.46 (62.8)
  C2D1 post-dose: number analyzed (Participants) | 2 | 4 | 0 | 35 | 30
  C2D1 post-dose | 2.86 (7.2) | 6.75 (42.2) |  | 8.31 (27.4) | 7.69 (38.3)
  C2D1 2 hrs post-dose: number analyzed (Participants) | 2 | 4 | 6 | 34 | 0
  C2D1 2 hrs post-dose | 2.38 (1.2) | 7.33 (44.7) | 7.65 (35.1) | 8.28 (26.7) |
  C2D2 pre-dose: number analyzed (Participants) | 0 | 0 | 6 | 0 | 0
  C2D2 pre-dose |  |  | 1.37 (38.6) |  |
  C2D2 post-dose: number analyzed (Participants) | 0 | 0 | 5 | 0 | 0
  C2D2 post-dose |  |  | 8.9 (34.1) |  |
  C3D1 pre-dose: number analyzed (Participants) | 3 | 4 | 5 | 33 | 8
  C3D1 pre-dose | 0.458 (36.3) | 1.08 (53.3) | 1.21 (45.1) | 1.11 (30.2) | 0.885 (43)
  C3D1 post-dose: number analyzed (Participants) | 3 | 4 | 5 | 34 | 26
  C3D1 post-dose | 3.37 (23.4) | 7.19 (30.8) | 6.66 (41.3) | 7.3 (39.2) | 6.76 (28.9)
  C4D1 pre-dose: number analyzed (Participants) | 3 | 4 | 4 | 32 | 32
  C4D1 pre-dose | 0.502 (36.9) | 1.09 (44.4) | 0.782 (90) | 1.03 (33.9) | 0.932 (52)
  C4D1 post-dose: number analyzed (Participants) | 3 | 4 | 4 | 32 | 28
  C4D1 post-dose | 3.24 (31.3) | 7.38 (26.3) | 4.09 (83) | 7.41 (44) | 5.55 (80.3)
  C5D1 pre-dose: number analyzed (Participants) | 3 | 4 | 3 | 30 | 4
  C5D1 pre-dose | 0.426 (51.7) | 1.02 (62) | 0.33 (176.6) | 1.12 (31.6) | 0.935 (106.1)

16. Secondary Outcome: Baseline Prevalence and Incidence of Treatment Emergent Anti-drug Antibodies (ADA) to Mosunetuzumab
Description: Participants are considered to have treatment-induced ADA responses if they are ADA negative or missing data at baseline and then develop an ADA response following study drug administration. Participants are considered to have treatment-enhanced ADA responses if they are ADA positive at baseline and the titer of one or more post baseline samples is at least 4-fold greater than the titer of the baseline sample. Patients are considered to be negative for ADAs if they are ADA negative at all timepoints or if they are ADA positive at baseline but do not have any post-baseline samples with a titer that is at least 4-fold greater than the titer of the baseline sample (treatment unaffected).
Time Frame: Cycles 1, 2, 6, 16, and at early discontinuation visit or at PRA (6-8 weeks after either C6D1 or last dose of study treatment)
Population: The immunogenicity analysis population included all participants with at least one ADA assessment. The number of participants analyzed are the values for baseline-evaluable participants and post-baseline evaluable participants.
Measure: Number; unit: Number of participants
Arm/Group | Group A1: Phase Ib Mosunetuzumab + CHOP | Group A2: Phase Ib Mosunetuzumab + CHOP | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized)
Number analyzed (Participants) | 3 | 4 | 8 | 40 | 38
Number of participants
  Positive sample at baseline: number analyzed (Participants) | 3 | 4 | 8 | 38 | 33
  Positive sample at baseline | 0 | 0 | 0 | 0 | 0
  Not positive at baseline: number analyzed (Participants) | 3 | 4 | 8 | 38 | 33
  Not positive at baseline | 3 | 4 | 8 | 38 | 33
  Positive for treatment-emergent ADA: number analyzed (Participants) | 3 | 4 | 6 | 39 | 37
  Positive for treatment-emergent ADA | 0 | 0 | 0 | 0 | 0
  Positive for treatment-induced ADA: number analyzed (Participants) | 3 | 4 | 6 | 39 | 37
  Positive for treatment-induced ADA | 0 | 0 | 0 | 0 | 0
  Positive for treatment-enhanced ADA: number analyzed (Participants) | 3 | 4 | 6 | 39 | 37
  Positive for treatment-enhanced ADA | 0 | 0 | 0 | 0 | 0
  Negative for treatment-emergent ADA: number analyzed (Participants) | 3 | 4 | 6 | 39 | 37
  Negative for treatment-emergent ADA | 3 | 4 | 6 | 39 | 37

17. Secondary Outcome: Baseline Prevalence and Incidence of Treatment Emergent ADA to Polatuzumab Vedotin
Description: as for outcome 16
Time Frame: Cycles 1, 2, 6, and at early discontinuation visit or at PRA (6-8 weeks after either C6D1 or last dose of study treatment)
Population: as for outcome 16
Measure: Number; unit: Number of participants
Arm/Group | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
Number analyzed (Participants) | 8 | 38 | 22
Number of participants
  Positive sample at baseline: number analyzed (Participants) | 8 | 38 | 21
  Positive sample at baseline | 0 | 1 | 2
  Not positive at baseline: number analyzed (Participants) | 8 | 38 | 21
  Not positive at baseline | 8 | 32 | 19
  Positive for treatment-emergent ADA: number analyzed (Participants) | 6 | 37 | 21
  Positive for treatment-emergent ADA | 0 | 0 | 1
  Positive for treatment-induced ADA: number analyzed (Participants) | 6 | 37 | 21
  Positive for treatment-induced ADA | 0 | 0 | 1
  Positive for treatment-enhanced ADA: number analyzed (Participants) | 6 | 37 | 21
  Positive for treatment-enhanced ADA | 0 | 0 | 0
  Negative for treatment-emergent ADA: number analyzed (Participants) | 6 | 37 | 21
  Negative for treatment-emergent ADA | 6 | 37 | 20

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months.
Description: All-cause mortality includes the entire population. Serious and non-serious adverse events are reported for the safety population, which consisted of all participants who received at least one dose of study drug, with participants grouped according to treatment received.
Arm/Group | Group A1: Phase Ib Mosunetuzumab + CHOP | Group A2: Phase Ib Mosunetuzumab + CHOP | Group B: Phase Ib Mosunetuzumab + CHP-Pola | Group C: Phase II Mosunetuzumab + CHOP | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized)
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/4 | 6/8 | 9/40 | 5/40 | 3/22
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/8 | 20/40 | 24/38 | 3/22
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 8/8 | 40/40 | 38/38 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A1: Phase Ib Mosunetuzumab + CHOP (N=3) | Group A2: Phase Ib Mosunetuzumab + CHOP (N=4) | Group B: Phase Ib Mosunetuzumab + CHP-Pola (N=8) | Group C: Phase II Mosunetuzumab + CHOP (N=40) | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) (N=38) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (7) | 5 (5) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A1: Phase Ib Mosunetuzumab + CHOP (N=3) | Group A2: Phase Ib Mosunetuzumab + CHOP (N=4) | Group B: Phase Ib Mosunetuzumab + CHP-Pola (N=8) | Group C: Phase II Mosunetuzumab + CHOP (N=40) | Arm 1: Phase II Mosunetuzumab + CHP-Pola (Randomized) (N=38) | Arm 2: Phase II Rituximab + CHP-Pola (Randomized) (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 2 (4) | 2 (4) | 17 (35) | 9 (13) | 5 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (6) | 19 (30) | 14 (24) | 7 (11)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (20) | 1 (1) | 3 (11) | 5 (6) | 6 (10) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4) | 5 (6) | 3 (3) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 8 (9) | 6 (6) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colonic haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 14 (17) | 6 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 12 (14) | 12 (17) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (7) | 22 (33) | 17 (24) | 9 (10)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (9) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (4) | 11 (18) | 9 (11) | 5 (7)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (2) | 0 (0) | 5 (5) | 1 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 5 (5) | 19 (23) | 12 (13) | 10 (13)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 2 (2) | 2 (3) | 8 (9) | 5 (7) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (6) | 8 (13) | 4 (4) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 24 (30) | 22 (27) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 3 (4) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 9 (10) | 2 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 10 (10) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 6 (6) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 2 (6)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (19) | 1 (3) | 3 (8)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 8 (13) | 11 (18) | 5 (7)
Platelet count decreased (Investigations) | 2 (4) | 1 (11) | 1 (1) | 5 (12) | 4 (8) | 3 (4)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 4 (4) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (10) | 6 (12) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 4 (4) | 15 (17) | 11 (13) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (3) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (14) | 2 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 5 (13) | 13 (25) | 4 (4) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (8) | 6 (6) | 4 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 2 (2) | 2 (9) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (12) | 4 (6) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 3 (3) | 2 (2) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (2)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 6 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 9 (14) | 2 (2) | 7 (8)
Horner's syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 13 (13) | 3 (3) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 5 (6) | 4 (4)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 2 (2) | 6 (6)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 7 (9) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 4 (4) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 12 (12) | 7 (7) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 6 (8) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 1 (1) | 9 (13) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03677141/Prot_SAP_000.pdf